CLINICAL TRIAL: NCT03628339
Title: Phase 1, Open-label, Single Sequence, Two-Period Crossover Trial to Evaluate the Effect of Tepotinib on CYP3A by Investigating the PK of the CYP3A Substrate Midazolam in Healthy Subjects
Brief Title: Effect of Tepotinib on PK of CYP3A Substrate Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: MS200095_0030; 2017-005055-92 (EudraCT Number)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Tepotinib; Midazolam; Cytochrome P450; Pharmacokinetics
MeSH Terms: interventions — Midazolam; tepotinib

STUDY DESIGN:
Intervention Model Description: This is a single sequence cross-over trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Reference Treatment) (Experimental): Participants received single oral dose of 7.5 milligrams (mg) midazolam tablet on Day 1 of treatment period 1. The washout period between midazolam administrations in Period 1 and Period 2 was 12 days.
  Interventions: Drug: Midazolam
- Tepotinib + Midazolam (Test Treatment) (Experimental): All participants who received 7.5 mg midazolam tablet in treatment period 1 received single oral dose of 500 mg tepotinib film-coated tablet from Day 1 to 11 along with 7.5 mg midazolam tablet on Day 11 in treatment period 2.
  Interventions: Drug: Midazolam; Drug: Tepotinib

INTERVENTIONS:
Drug: Midazolam — Participant received single oral dose of 7.5 mg midazolam tablet on Day 1 of treatment period 1 and Day 11 in treatment period 2.
Drug: Tepotinib — Participants received single oral dose of 500 mg tepotinib film-coated tablet from Day 1 to 11 in treatment period 2.
  Arms: Tepotinib + Midazolam (Test Treatment)

SUMMARY:
The study investigated the effect of tepotinib on the pharmacokinetics (PK) of the Cytochrome P450 (CYP) 3A substrate midazolam determined from concentrations of midazolam and its main metabolite 1-hydroxymidazolam in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-child bearing potential
* Body weight between 50 to 100 kilogram (kg)
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical study within 60 days prior to first drug administration
* Whole blood donation or loss of greater than 450 milliliter (mL) within 60 days prior to first drug administration
* Any surgical or medical condition, or any other significant disease that could interfere with the study objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

REFERENCES:
- [Derived] Yalkinoglu O, Becker A, Krebs-Brown A, Vetter C, Lupfert C, Perrin D, Heuer J, Biedert H, Hirt S, Bytyqi A, Bachmann A, Strotmann R. Assessment of the potential of the MET inhibitor tepotinib to affect the pharmacokinetics of CYP3A4 and P-gp substrates. Invest New Drugs. 2023 Aug;41(4):596-605. doi: 10.1007/s10637-023-01378-z. Epub 2023 Jul 6. PMID 37415001
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0030
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 25 participants were screened in this study. Out of which, 12 participants received Midazolam and Tepotinib + Midazolam treatment.
Period: Treatment Period 1
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Started | 0 | 12
Completed | 0 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who received single oral dose of 7.5 mg midazolam tablet on Day 1 of treatment period 1 and oral dose of 500 mg tepotinib film-coated tablet from Day 1 to 11 along with 7.5 mg midazolam tablet on Day 11 in treatment period 2. The washout period between midazolam administrations in Period 1 and Period 2 was 12 days.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to Last Sampling Time (Tlast) at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Midazolam
Description: AUC0-t a Pharmacokinetic (PK) parameter was calculated according to the mixed log linear trapezoidal rule.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 and 43 hours post-dose on Day 1 of period 1 and Day 11 of Period 2
Population: PK Analysis Set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results, who have received at least one dose of midazolam and who have at least 3 post-dose concentration measurements.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*picogram per milliliter (h*pg/mL)
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
hour*picogram per milliliter (h*pg/mL) | 107969 (42.0) | 109477 (46.5)
Statistical Analysis 1: Comparison: Midazolam (Reference Treatment) vs Tepotinib + Midazolam (Test Treatment); Test type: Other; % Ratio of Geometric Least square Mean = 101.40, 90% CI 2-sided [89.35 to 115.06]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Midazolam
Description: AUC0-inf was calculated as AUC0-t plus (+) AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastpred/Lambda z, where Clastpred is the predicted plasma concentration at the last sampling time point, calculated from the log-linear regression line for Lambda z determination at which the measured plasma concentration is at or above Lower limit of quantification (LLOQ).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
h*pg/mL | 109285 (41.9) | 110550 (46.2)
Statistical Analysis 1: Comparison: Midazolam (Reference Treatment) vs Tepotinib + Midazolam (Test Treatment); Test type: Other; % Ratio of Geometric Least square Mean = 101.16, 90% CI 2-sided [89.24 to 114.66]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam
Description: Cmax was obtained directly from concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
pg/mL | 49172 (59.7) | 50954 (54.1)
Statistical Analysis 1: Comparison: Midazolam (Reference Treatment) vs Tepotinib + Midazolam (Test Treatment); Test type: Other; % Ratio of Geometric Least square Mean = 103.62, 90% CI 2-sided [86.91 to 123.56]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Midazolam and Midazolam Metabolite (1-Hydroxymidazolam)
Description: Tmax is time to reach maximum observed plasma concentration obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Hours
  Midazolam | 0.500 [0.500 to 1.50] | 0.508 [0.483 to 2.00]
  Midazolam Metabolite (1- Hydroxymidazolam) | 0.500 [0.500 to 2.00] | 0.508 [0.483 to 2.00]

5. Secondary Outcome: Elimination Half Life (t1/2) of Midazolam and Midazolam Metabolite (1-Hydroxymidazolam)
Description: Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Hours
  Midazolam | 5.52 (31.4) | 4.81 (41.2)
  Midazolam Metabolite (1- Hydroxymidazolam) | 6.34 (29.8) | 6.90 (26.8)

6. Secondary Outcome: Area Under Plasma Concentration-time Curve From Time Zero to Last Sampling Time (Tlast) at Which the Concentration is at or Above the Lower Limit of Quantification (AUC0-t) of Midazolam Metabolite (1-Hydroxymidazolam)
Description: AUC0-t a Pharmacokinetic (PK) parameter was calculated according to the mixed log linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
h*pg/mL | 30589 (23.8) | 32627 (25.1)

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Midazolam Metabolite (1-Hydroxymidazolam)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*pg/mL
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
h*pg/mL | 31269 (23.0) | 33372 (24.4)

8. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Midazolam Metabolite (1-Hydroxymidazolam)
Description: Cmax was obtained directly from concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
pg/mL | 14909 (60.4) | 15852 (34.7)

9. Secondary Outcome: Metabolic Ratio of Midazolam and Midazolam Metabolite (1-hydroxymidazolam)
Description: Metabolic ratio was calculated as AUC 0-infinity of midazolam divided by AUC 0-infinity of 1-hydroxymidazolam.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
ratio | 0.286 (37.2) | 0.302 (34.3)

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Death
Description: Adverse event (AE) was defined as any untoward medical occurrence in participants which does not necessarily have causal relationship with treatment. AE was any unfavorable and unintended sign (including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. A serious adverse event (SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Baseline (Day 1 of treatment period 1) up to the End of Trial visit (Day 20)
Population: Safety Analysis Set included all participants who have received atleast 1 dose of planned investigational medicinal product (IMP). Participants was analyzed according to the actual treatment they receive.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Participants
  TEAEs | 1 | 10
  Serious TEAEs | 0 | 0
  TEAEs Leading to Death | 0 | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Values
Description: Number of participants with clinically significant changes in laboratory values were reported. Clinical significance was decided by the investigator. Laboratory investigation included hematology and urinalysis.
Time Frame: From Screening up to the End of Trial visit (Day 20)
Population: Safety Analysis Set included all participants who have received atleast 1 dose of planned IMP. Participants was analyzed according to the actual treatment they receive.
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in 12-Lead Electrocardiogram (ECG)
Description: Number of participants with clinically significant changes in 12-lead ECG were reported. Clinical significance was decided by the investigator. The 12-lead ECGs were recorded after the participants have rested for at least 5 minute in supine position.
Time Frame: Day 1 (Treatment Period 1) up to the End of Trial visit (Day 20)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant changes in vital signs were reported. Clinical significance was decided by Investigator. Vital signs included body temperature, blood pressure and pulse rate.
Time Frame: Day 1 (Treatment Period 1) up to the End of Trial visit (Day 20)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline (Day 1 of treatment period 1) up to the End of Trial visit (Day 20)
Arm/Group | Midazolam (Reference Treatment) | Tepotinib + Midazolam (Test Treatment)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Midazolam (Reference Treatment) (N=12) | Tepotinib + Midazolam (Test Treatment) (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 4
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Medical device site reaction (General disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-06-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03628339/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT03628339/SAP_001.pdf